CLINICAL TRIAL: NCT04157088
Title: A Randomized, Open-label, Multicenter, Phase 2b Study to Evaluate Physical Function, Including Balance and Daily Activity, in Participants With Castration-resistant Prostate Cancer Treated With Darolutamide or Enzalutamide
Brief Title: Study to Compare the Effects of Drug Darolutamide and Drug Enzalutamide on Physical Function, Including Balance and Daily Activity, in Patients With Castration-resistant Prostate Cancer (CRPC)
Acronym: DaroAcT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The results of the lead-in phase did not fulfill the criteria set for moving into the randomized phase
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20609
Record Dates: First submitted 2019-10-21; First posted 2019-11-08 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Prostatic Cancer, Castration-Resistant
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — darolutamide; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants treated with darolutamide (Experimental)
  Interventions: Drug: Darolutamide (Nubeqa, BAY1841788)
- Participants treated with enzalutamide (Experimental)
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Darolutamide (Nubeqa, BAY1841788) — 600mg, twice daily
  Arms: Participants treated with darolutamide
Drug: Enzalutamide — 160mg, once daily
  Arms: Participants treated with enzalutamide

SUMMARY:
Researchers in this study want to compare the effects of drug darolutamide and drug enzalutamide on physical function, including balance and daily activity, in patients with castration-resistant prostate cancer (CRPC). Both darolutamide and enzalutamide are approved AR inhibitors used for the treatment of patients with CRPC. AR inhibitor is a substance that keeps androgens (male sex hormones) from binding to proteins called androgen receptors, which are found in normal prostate cells, some prostate cancer cells, and in some other cells. Preventing this binding blocks the effects of these hormones in the body and therefore keeps prostate cancer cells from growing. Patients participating this study will receive either darolutamide or enzalutamide tablets. To evaluate the physical function, patients will be asked to make some movements like rising from a chair, walking three meters, etc. Additionally, researchers also want to find out the survival of patients and if patients have fatigue (feeling tired), cognitive (learning and thinking) problems, or other medical problems during the trial. Brand name of darolutamide is Nubeqa; brand name of enzalutamide is Xtandi.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age inclusive or older at the time of signing the informed consent.
* Participants who have:

  * Histologically or cytologically confirmed adenocarcinoma of prostate, CRPC (Castration-resistant prostate cancer) defined by disease progression despite ADT (Androgen deprivation therapy) and may present as either a confirmed rise in serum PSA (Prostate-specific antigen) levels (as defined by PCWG3 (Prostate Cancer Working Group)), the progression of pre-existing disease, and/or the appearance of new metastases. Metastatic and non-metastatic CRPC patients will be eligible.
  * KPS (Karnofsky Performance Scale) performance status of ≥80
  * Blood counts at screening: hemoglobin ≥9.0 g/dL, absolute neutrophil count ≥1500/μL, platelet count ≥100,000/μL
  * Screening values of serum alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤2.5 × upper limit of normal (ULN), total bilirubin ≤1.5 × ULN, creatinine ≤2.0 × ULN
  * Life expectancy of at least 1 year
* Sex: Male

Exclusion Criteria:

* Symptomatic local-regional disease that requires medical intervention including moderate/severe urinary obstruction or hydronephrosis with abnormal renal function due to prostate cancer. Participants with visceral metastasis will be excluded.
* Past (within 6 months before the start of study intervention) or concurrent stroke, myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, and/or congestive heart failure (New York Heart Association Class III or IV)
* Prior malignancy. Adequately treated basal cell or squamous cell carcinoma of the skin or superficial bladder cancer that has not spread behind the connective tissue layer (i.e. pTis, pTa, and pT1) is allowed, as well as any other cancer for which treatment has been completed 3 years before the start of study intervention and from which the participant has been disease free
* Prior or concurrent central nervous system disease, such as epilepsy, Parkinson's disease, Alzheimer's disease, dementia, or multiple sclerosis
* Non-ambulatory participants who need a wheelchair. Other assistive devices (e.g., cane or walker) are permitted.
* Clinically significant limitations in cognitive function and/or physical function, such as >20 seconds in the TUG assessment
* Prior treatment with any of the following:

  * Second-generation AR inhibitors, such as enzalutamide, apalutamide, or Darolutamide
  * Other investigational AR inhibitors
  * Progression on abiraterone acetate and discontinuation within 6 months before signing the ICF for the study
  * For mCRPC participants: any chemotherapy, and/or >2 prior lines of systemic anticancer treatment. Treatment with an LHRH agonist, LHRH antagonists, or orchidectomy is not counted as systemic treatment with regard to this exclusion criterion.
* Use of immunotherapy within 28 days before the start of study intervention
* Treatment with radiotherapy/radiopharmaceuticals within 12 weeks before the start of study intervention
* Previous participation in other clinical studies within 28 days before the start of study treatment or 5 half-lives of the investigational treatment of the previous study, whichever is longer Diagnostic assessments

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Oregon Health and Science University, Portland, Maine
  - New Jersey Urology, LLC, Voorhees Township, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - MidLantic Urology - Bala Cynwyd, Bala-Cynwyd, Pennsylvania
  - Bon Secours St. Francis Hospital, Greenville, South Carolina
  - Carolina Urological Research Center, Myrtle Beach, South Carolina

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 centers in United States of America (USA) between 17 Dec 2019 (First participant first visit) and 08 JUL 2022 (Last participant last visit).
Pre-assignment Details: 40 participants were screened into the study (signed informed consent form (ICF)). 10 participants failed screening as they did not meet the inclusion/exclusion criteria. None of these patients received treatment. 30 participants were enrolled in the study, all 30 participants only received the darolutamide treatment during the lead-in phase as the study was terminated prior to the initiation of the randomized phase.
Groups:
- Participants Treated With Darolutamide: Participants treated with darolutamide 600 mg (2 tablets of 300 mg) twice daily with food, equal to a total daily dose of 1200 mg.
Period: Overall Study
Arm/Group | Participants Treated With Darolutamide
Started | 30
Received Treatment | 30
Participants Off-Study | 30
Completed | 0
Not Completed | 30
Not completed — Study terminated by sponsor | 23
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (8.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 14
  More than one race | 0
  Unknown or Not Reported | 9
Short Physical Performance Battery (SPPB) [Mean (Standard Deviation); unit: units on a scale] — The SPPB is a group of measures that combines the results of the gait speed, chair stand and balance tests. The composite SPPB score ranges from 0 (worst performance) to 12 (best performance)
  units on a scale | 8.17 (1.577)
Counts per minute (CPM) [Mean (Standard Deviation); unit: Mean count per minute] — Participants required at least 2 valid days to be included in the analysis at each visit. 'Valid' is defined as at least 10 awake wear hours. CPM for each valid day is defined as 'awake wear-filtered total vector magnitude counts' divided by 'awake wear minutes'. Population: The number of all enrolled participants is n=30. The full analysis set FAS considers all enrolled participants who signed the ICF, n=30. The safety analysis set SAF considers all enrolled participants that have actually received an intervention. Of 30 participants, 27 received this intervention.
  Mean count per minute
    number analyzed (Participants) | 27
    (all) | 1900.4 (448.442)
Cognitive function: Hopkins Verbal Learning Test Revised (HVLT-R) [Mean (Standard Deviation); unit: units on a scale] — The HVLT-R is a learning and memory test, in which the participant is asked to learn and recall a list of 12 words over three trials.
  The HVLT-R TR (total score) score ranges from 0 to 36, where higher scores indicated greater verbal learning and recall.
  The HVLT-R DR (delayed recall) score ranges from 0 to 12, where higher scores indicated greater verbal learning and recall.
  The HVLT-R RECOG (Delayed Recognition) score ranges from -12 to 12, where higher scores indicated better performance. Population: The number of all enrolled participants is n=30. The full analysis set FAS considers all enrolled participants who signed the ICF, n=30. The safety analysis set SAF considers all enrolled participants that have actually received an intervention. Of 30 participants, 29 received the HVLT-R DR and HVLT-R RECOG interventions.
  units on a scale
    HVLT-R TR | 19.2 (6.24)
    HVLT-R DR: number analyzed (Participants) | 29
    HVLT-R DR | 7.1 (3.14)
    HVLT-R RECOG: number analyzed (Participants) | 29
    HVLT-R RECOG | 9.1 (2.48)
Cognitive function: Trail Making Test (TMT) [Mean (Standard Deviation); unit: seconds] — TMT Part A (TMTA) is timed up to a maximum of 3 minutes, and TMT Part B (TMTB) is timed up to a maximum of 5 minutes. The lower score indicated the better performance. Population: The number of all enrolled participants is n=30. The full analysis set FAS considers all enrolled participants who signed the ICF, n=30. The safety analysis set SAF considers all enrolled participants that have actually received an intervention. Of 30 participants, 30 performed the TMTA intervention, 29 received the TMTB intervention.
  seconds
    TMTA | 50.4 (31.46)
    TMTB: number analyzed (Participants) | 29
    TMTB | 113.0 (64.17)
Cognitive function: Controlled Oral Word Association (COWA) [Mean (Standard Deviation); unit: units on a scale] — The COWA test assessed lexical fluency. Given a specific letter of the alphabet, participants were required to produce as many words as possible that begin with that letter. There were two alternate forms of the COWA, each with three unique letter exemplars. The lowest possible score is zero, meaning no words could be produced. There is no limit to the higher end of the scale given that participants can produce as many words as possible for each of the three letters. Higher scores indicate greater word retrieval and better cognitive function.
  units on a scale | 31.7 (13.87)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Worsening in TUG Time During the 24- Week Period.
Description: TUG: Timed Up & Go. Worsening is defined as an increase of at least 1 second in TUG time from baseline. (The minimum clinically important difference [MCID] in TUG time is 1 second
Time Frame: Up to 24 weeks
Population: Full analysis set: All enrolled participants (30). 2 participants were excluded from analysis due to screening assessment performed in 4 meters instead of 3 meters.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 28
Participants
  At week 12: number analyzed (Participants) | 22
  At week 12 | 5
  At week 24: number analyzed (Participants) | 23
  At week 24 | 5
  During the 24-week period: number analyzed (Participants) | 25
  During the 24-week period | 8

2. Secondary Outcome: Number of Participants With an Increase of at Least 1 Second in TUG Time at 12 and 24 Weeks and During the 52 Weeks.
Description: Worsening was defined as an increase of at least 1 second in TUG time from baseline.
  Improved was defined at least 1 second decrease from baseline. Stable was defined as change from baseline between less than 1 second increase and less than 1 second decrease.
Time Frame: At 12 week, 24 week and 52 week.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 28
Participants
  At week 12_Stable: number analyzed (Participants) | 22
  At week 12_Stable | 15
  At week 12_Worsen: number analyzed (Participants) | 22
  At week 12_Worsen | 5
  At week 12_ Improved: number analyzed (Participants) | 22
  At week 12_ Improved | 2
  At week 24_Stable: number analyzed (Participants) | 23
  At week 24_Stable | 17
  At week 24_Worsen: number analyzed (Participants) | 23
  At week 24_Worsen | 5
  At week 24_ Improved: number analyzed (Participants) | 23
  At week 24_ Improved | 1
  At week 52_Stable: number analyzed (Participants) | 19
  At week 52_Stable | 14
  At week 52_Worsen: number analyzed (Participants) | 19
  At week 52_Worsen | 5
  At week 52_ Improved: number analyzed (Participants) | 19
  At week 52_ Improved | 0

3. Secondary Outcome: Time to Worsening (Increase of at Least 1 Second) in TUG Time
Description: At the end of the lead-in phase, the overall feasibility of the study execution was assessed and decided not to proceed with the randomized phase. Therefore, data on this outcome which needed to be collected in the randomized phase was unavailable.
Time Frame: From randomization to the first date a participant had a worsening.
Population: At the end of the lead-in phase, the overall feasibility of the study execution was assessed and decided not to proceed with the randomized phase. Therefore, data on this outcome which needed to be collected in the randomized phase was unavailable.
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With a Worsening in SPPB Total Score at 12 and 24 Weeks and During the 24 Weeks and 52 Weeks From Baseline.
Description: The SPPB is a group of measures that combines the results of the gait speed, chair stand and balance tests. The composite SPPB score ranges from 0 (worst performance) to 12 (best performance)
Time Frame: At 12 and 24 weeks and during the 24 weeks and 52 weeks from baseline
Population: Full analysis set: All enrolled participants (30).
  1 participant at week 24 visit was excluded from analysis due to being performed outside of visit window.
Measure: Number; unit: Participants
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 30
Participants
  At week 12: number analyzed (Participants) | 22
  At week 12 | 3
  At week 24: number analyzed (Participants) | 24
  At week 24 | 8
  At week 52: number analyzed (Participants) | 22
  At week 52 | 7

5. Secondary Outcome: Mean Change From Baseline in Daily Physical Activity as Assessed by CPM, at 12 and 24 Weeks, and During the 24 Weeks and 52 Weeks From Baseline.
Description: Participants required at least 2 valid days to be included in the analysis at each visit. 'Valid' is defined as at least 10 awake wear hours. CPM for each valid day is defined as 'awake wear-filtered total vector magnitude counts' divided by 'awake wear minutes''. A participant's CPM at each visit is the average of daily CPM.
Time Frame: At 12 week, 24 week and 52 week
Population: Safety Analysis Set: All enrolled participants who received any quantity of study intervention, regardless of their eligibility for the study.
Measure: Mean (Standard Deviation); unit: Mean counts per minute
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 30
Mean counts per minute
  At week 12: number analyzed (Participants) | 20
  At week 12 | 60.04 (266.480)
  At week 24: number analyzed (Participants) | 19
  At week 24 | 83.74 (455.580)
  At week 52: number analyzed (Participants) | 14
  At week 52 | -37.73 (304.621)

6. Secondary Outcome: Mean Change From Baseline in Accelerometer-assessed Proportion of Time Spent in Light to Vigorous Physical Activity Based on a Threshold of >100 Activity Counts Per Minute.
Description: as for outcome 3
Time Frame: At 12, 24, and 52 weeks for the randomization phase
Population: as for outcome 3
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With a Decline in Cognitive Function During the 24 Weeks and 52 Weeks From Baseline, as Assessed by HVLT-R.
Description: The HVLT-R is a learning and memory test, in which the participant is asked to learn and recall a list of 12 words over three trials. The HVLT-R TR (total score) score ranges from 0 to 36, where higher scores indicated greater verbal learning and recall. The HVLT-R DR (delayed recall) score ranges from 0 to 12, where higher scores indicated greater verbal learning and recall. The HVLT-R RECOG (Delayed Recognition) score ranges from -12 to 12, where higher scores indicated better performance.
Time Frame: During the 24 weeks and 52 weeks from baseline.
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 30
Participants
  HVLT-R TR_At week 24: number analyzed (Participants) | 26
  HVLT-R TR_At week 24 | 5
  HVLT-R TR_At week 52: number analyzed (Participants) | 22
  HVLT-R TR_At week 52 | 5
  HVLT-R DR_At week 24: number analyzed (Participants) | 25
  HVLT-R DR_At week 24 | 4
  HVLT-R DR_At week 52: number analyzed (Participants) | 21
  HVLT-R DR_At week 52 | 3
  HVLT-R RECOG_At week 24: number analyzed (Participants) | 25
  HVLT-R RECOG_At week 24 | 5
  HVLT-R RECOG_At week 52: number analyzed (Participants) | 21
  HVLT-R RECOG_At week 52 | 3

8. Secondary Outcome: Number of Participants With a Decline in Cognitive Function During the 24 Weeks and 52 Weeks From Baseline, as Assessed by TMT.
Description: TMT Part A (TMTA) is timed up to a maximum of 3 minutes, and TMT Part B (TMTB) is timed up to a maximum of 5 minutes. The lower score indicated the better performance.
Time Frame: During the 24 weeks and 52 weeks from baseline.
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 30
Participants
  TMTA_At week 24: number analyzed (Participants) | 26
  TMTA_At week 24 | 5
  TMTA_At week 52: number analyzed (Participants) | 22
  TMTA_At week 52 | 3
  TMTB_At week 24: number analyzed (Participants) | 23
  TMTB_At week 24 | 6
  TMTB_At week 52: number analyzed (Participants) | 19
  TMTB_At week 52 | 4

9. Secondary Outcome: Number of Participants With a Decline in Cognitive Function During the 24 Weeks and 52 Weeks From Baseline, as Assessed by COWA.
Description: The COWA test assessed lexical fluency. Given a specific letter of the alphabet, participants were required to produce as many words as possible that begin with that letter. There were two alternate forms of the COWA, each with three unique letter exemplars. The lowest possible score is zero, meaning no words could be produced. There is no limit to the higher end of the scale given that participants can produce as many words as possible for each of the three letters. Higher scores indicate greater word retrieval and better cognitive function.
Time Frame: During the 24 weeks and 52 weeks from baseline.
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 30
Participants
  At week 24: number analyzed (Participants) | 26
  At week 24 | 3
  At week 52: number analyzed (Participants) | 22
  At week 52 | 2

10. Secondary Outcome: Number of Participants With a Decline Using a Selected Domain of Functional Assessment of Cancer Therapy-Cognitive (FACT-Cog).
Description: FACT-Cog with a range of 0-28 points, higher score is better. Decline was defined as a decrease of >10 points during the 24 weeks and 52 weeks from baseline.
Time Frame: During the 24 weeks and 52 weeks from baseline.
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 30
Participants
  During the 24-week period: number analyzed (Participants) | 24
  During the 24-week period | 0
  During the 52-week period: number analyzed (Participants) | 25
  During the 52-week period | 3

11. Secondary Outcome: Number of Participants With a Worsening of Fatigue During the 24 Weeks and 52 Weeks.
Description: as for outcome 3
Time Frame: Up to 52 weeks in randomization phase.
Population: as for outcome 3
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With an Increase of at Least 1 Point in Fatigue Interference by 24 Weeks and 52 Weeks From Baseline (Based on Items 4A-F of the BFI)
Description: Fatigue Interference decline is defined as an increase of at least 1 point in any Fatigue Interference from baseline.
  BFI: Brief Fatigue Inventory. BFI is a 5 minute self-assessment tool that identifies fatigue in cancer participants over a 24-hour period.
Time Frame: At 24 weeks and 52 weeks
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 30
Participants
  During the 12 week period: number analyzed (Participants) | 29
  During the 12 week period | 10 [17.9 to 54.3]
  During the 24 week period: number analyzed (Participants) | 29
  During the 24 week period | 12 [23.5 to 61.1]
  During the 52 week period: number analyzed (Participants) | 29
  During the 52 week period | 13 [26.4 to 64.3]

13. Secondary Outcome: Number of Participants With a Worsening in Scores in the PHQ-9 During the 24 Weeks and 52 Weeks From Baseline.
Description: as for outcome 3
Time Frame: Up to 52 weeks in randomization phase
Population: as for outcome 3
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Participants With Treatment Emergent AEs, SAEs, and AEs Leading to Study Intervention Discontinuation
Description: Treatment-Emergent Adverse Events (TEAEs) were defined as any events arising or worsening after the first dose of study drug until 30 days after last dose.
  SAEs: Serious adverse events
Time Frame: Up to 52 weeks
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 30
Participants
  TEAEs | 26
  SAEs | 6
  AEs leading to study intervention discontinuation | 3

15. Secondary Outcome: Number of Participants With AEs of Interest, Including Falls, Fractures, and Hypothyroidism
Description: AEs of interest were followed up regardless of causality or relationship to study intervention.
Time Frame: Up to 52 weeks
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 30
Participants
  Falls | 1
  Fractures | 1
  Hypothyroidism | 0

16. Secondary Outcome: Time to Deterioration of Karnofsky Performance Scale (KPS) Defined as at Least a 10 Point Decline From Baseline.
Description: as for outcome 3
Time Frame: From randomization to the first date the participant had had a decline in KPS of at least 10 points.
Population: as for outcome 3
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 0

17. Secondary Outcome: Number of Participants With Treatment Exposure of the Study Intervention Including Time on Treatment
Description: A total of 30 participants received treatment with darolutamide 600 mg twice daily in the lead-in phase of the study, comprising the safety evaluable population.
  No participant received either darolutamide or enzalutamide in the randomized phase of the study as the study was terminated prematurely prior to the initiation of the randomized phase of the study.
Time Frame: Up to 52 weeks
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 30
Participants | 30

18. Secondary Outcome: Number of Participants With Dose Reductions of Study Intervention
Description: as for outcome 3
Time Frame: Up to 52 weeks in randomization phase
Population: as for outcome 3
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 0

19. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression (as Per Prostate Cancer Working Group [PCWG3] Criteria)
Description: as for outcome 3
Time Frame: From randomization to the time when the criteria for PSA progression (according to PCWG3) was met, up to 52 weeks.
Population: as for outcome 3
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 0

20. Secondary Outcome: Survival Status
Description: as for outcome 3
Time Frame: Up to 52 weeks in randomization phase
Population: as for outcome 3
Arm/Group | Participants Treated With Darolutamide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Timeframe for TEAEs: after the first dose of study drug until 30 days after last dose, with a maximum duration of 815 days. Timeframe for the all-cause mortality: All deaths that occurred at any time during the study before the last contact, with a maximum duration of 847 days.
Arm/Group | Participants Treated With Darolutamide
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 6/30
Other Adverse Events (participants affected / at risk) | 21/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Treated With Darolutamide (N=30)
Cardiac failure (Cardiac disorders) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Treated With Darolutamide (N=30)
Constipation (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 8 (8)
Oedema peripheral (General disorders) | 2 (3)
COVID-19 (Infections and infestations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Dizziness (Nervous system disorders) | 4 (4)
Haematuria (Renal and urinary disorders) | 5 (5)
Pollakiuria (Renal and urinary disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Hypertension (Vascular disorders) | 2 (4)
Hypotension (Vascular disorders) | 2 (2)
Hot flush (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
A total of 30 participants received treatment with darolutamide 600 mg twice daily in the lead in phase of the study, comprising the safety evaluable population.

No participant received either darolutamide or enzalutamide in the randomized phase of the study as the study was terminated prematurely prior to the initiation of the randomized phase of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT04157088/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/88/NCT04157088/SAP_001.pdf